CLINICAL TRIAL: NCT05134844
Title: Comparison of the Effect of Halliwick Hydrotherapy in Snoezelen Multisensory Environment and Snoezelen Intervention in Children With Autism
Brief Title: Halliwick Hydrotherapy and Snoezelen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantinos Chandolias, Post doc researcher Dr Konstantinos Chandolias, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36469
Record Dates: First submitted 2021-11-11; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Autism Spectrum Disorder; Autism; Sensory Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Sensation Disorders

STUDY DESIGN:
Intervention Model Description: The design of the present study included two groups of children with autism. A first group of 26 children formed the core group with the Halliwick philosophy - hydrotherapy in water in a multi-sensory Snoezelen environment. A second group of 27 children was the Snoezelen on-site control-intervention group with two sessions per week, which was the measure of comparison and support of "reasonable" hypotheses, in order to evaluate the hypothesis that Halliwick hydrotherapy in a multi-sensory environment in combination with intervention on land leads to better therapeutic results.
  The application of the tests was done by the 2 examiners, who were pediatric physiotherapists - hydrotherapists with many years of experience (more than 10 years) in approaching motor problems of children with stroke. The tests were videotaped and then graded by the two examiners separately, which was considered important in order to ensure the objective grading of the assessment tests.
Who Masked: Participant
Masking Description: A first group of 26 children formed the core group with the Halliwick philosophy - hydrotherapy in water in a multi-sensory Snoezelen environment. A second group of 27 children was the Snoezelen on-site control-intervention group with two sessions per week,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Halliwick Snoezelen Group (Experimental): Hydrotherapy in a multi-sensory Snoezelen environment
  Interventions: Other: Hydrotherapy- Snoezelen; Other: Snoezelen
- Land Snoezelen Group (Experimental): Land multi-sensory Snoezelen environment
  Interventions: Other: Hydrotherapy- Snoezelen; Other: Snoezelen

INTERVENTIONS:
Other: Hydrotherapy- Snoezelen — Multi sensory approach in water
Other: Snoezelen — Multu Sensory approach on land

SUMMARY:
The aim of this study was to evaluate the effectiveness of the Halliwick concept in the adapted Snoezelen multi-sensory environment, in the gross mobility of children belonging to the autism spectrum.

DETAILED DESCRIPTION:
The study involved 54 children, aged 4 to 8, all of whom belonged to the autism spectrum (ASD) and all had cognitive limitations. The duration of the intervention was 3 months by specialized pediatric physiotherapists and hydrotherapists certified by the program "PEDIATRIC SPECIALIZATION" and NDT- BOBATH. All children were assessed through the WOTA 1 and PEDI assessment tests.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-8 years with autism
* All participants had the criterion of participation in the monitoring treatment program by the same therapist either in water or on land.

Exclusion Criteria:

* Children with other neurological diseases were excluded.
* Children who had some scheduled surgery were also excluded intervention or injection of sausage toxin.
* Children who were absent from the treatment program were excluded either in water or on land for more than a week.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Disability and Activity- PEDI | 3 months
  Pediatric Evaluation of Disability Inventory assesses key functional capabilities and performance in children ages 6 months to 7 years. PEDI is also useful for older children whose functional abilities are lower than those of seven-year-olds without disabilities.
Adaptation and progression in pool- WOTA | 3 months
  Water Orientation test Alyn- Wota is an assessment scale to evaluate the progress of a patient in the water enviroment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamía, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Ager, A., & O'May, F. (2001). Issues in the definition and implementation of ''best practice'' for staff delivery of interventions for challenging behaviour. Journal of Intellectual & Developmental Disability, 26, 243-256. 2. American Academy of Child and Adolescent Psychiatry. Practice Parameters for the assessment and treatment of Children, Adolescents and Adults with Autism and Other Pervasive Developmental Disorders. 1999, 38(12) Supplement, 32S-54S. 3. American Psychiatric Association. Autism spectrum disorder. In: Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, American Psychiatric Association, Arlington, VA 2013. p.50 4. American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders,4th edition(DSM-IV).Washington, DC 1994: American Psychiatric Association. 5. Anderson GM, Hoshiono Y. Neurochemical studies of autism. In: Cohen DJ, Volkmar FR (eds) Handbook of Autism and Pervasive Developmental Disorders. New York: Wiley, 1997, pp. 325-343. 6. Ashby, M., Broxholme, S., Pitcaithly, D., & Lindsay, W. R. (1995). Snoezelen: Its effects on concentration and responsiveness in people with profound multiple handicaps. British Journal of Occupational Therapy, 58, 303-307. 7. Atari, R. (2014). The Influence of Multi-Sensory Environment on Physiological Response in Children with Autism Spectrum Disorders and Children with Special Health Care Needs. Marquette University. 8. Bailey A & Lord C. Autism Spectrum Disorder. In M. Rutter & E. Taylor (eds) Child and Adolescent Psychiatry 4th Edition. Oxford: Blackwell Publishing 2002, pp. 636-663. 9. Bailey A, Le Couteur A, Gottesman I et al. Autism as a strongly genetic disorder: evidence from a British twin study. Psychological Medicine, 1995, 25: 63-77. 10. Bailey A, Palferman S, Heavey L, Le Couteur A. Autism: the phenotype in relatives. Journal of Autism and Developmental Disorders, 1998, 28(5): 369-392.